CLINICAL TRIAL: NCT02154347
Title: Post-marketing Clinical Trial of KAD-1229 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KAD6401
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mitiglinide; Insulin

ARMS (2):
- KAD-1229/KAD-1229 (Experimental): Patients are administered KAD-1229 for 16 weeks (double-blind period), followed by KAD-1229 for up to 52 weeks (open-label period) with insulin throughout the study.
  Interventions: Drug: KAD-1229; Drug: Insulin
- Placebo/KAD-1229 (Other): Patients are administered Placebo for 16 weeks (double-blind period), followed by KAD-1229 for up to 52 weeks (open-label period) with Insulin throughout the study.
  Interventions: Drug: KAD-1229; Drug: Placebo; Drug: Insulin

INTERVENTIONS:
Drug: KAD-1229
Drug: Placebo
  Arms: Placebo/KAD-1229
Drug: Insulin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of KAD-1229 as combination therapy with insulin for 16 weeks and up to 52 weeks administration in patients with type 2 Diabetes Mellitus who show inadequate glycemic control with diet, and insulin monotherapy, or insulin and oral hypoglycemic agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has been receiving dietary therapy and a stable dose and regimen of insulin over 8 weeks before at the time of an observation term start
* Patients whose HbA1c at the time of an observation term start is 7.5% or more and less than 10.0%

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Patients with serious diabetic complications and other serious complications

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Primary Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/KAD-1229: Patients are administered Placebo for 16 weeks (double-blind period), followed by KAD-1229 for up to 52 weeks (open-label period) with Insulin throughout the study.
  KAD-1229
  Placebo
  Insulin
- KAD-1229/KAD-1229: Patients are administered KAD-1229 for 16 weeks (double-blind period), followed by KAD-1229 for up to 52 weeks (open-label period) with insulin throughout the study.
  KAD-1229
  Insulin
Period: Double-blind Period
Arm/Group | Placebo/KAD-1229 | KAD-1229/KAD-1229
Started | 60 | 118
Completed | 57 | 114
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Open-label Period
Arm/Group | Placebo/KAD-1229 | KAD-1229/KAD-1229
Started | 57 | 113
Completed | 50 | 88
Not Completed | 7 | 25
Not completed — Adverse Event | 3 | 4
Not completed — Lack of Efficacy | 4 | 19
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/KAD-1229 | KAD-1229/KAD-1229 | Total
Number analyzed (Participants) | 60 | 118 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.7) | 59.7 (10.3) | 58.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 39 | 48
  Male | 51 | 79 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 60 | 118 | 178
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HbA1c [Mean (Standard Deviation); unit: %] | 8.54 (0.85) | 8.48 (0.70) | 8.50 (0.75)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c
Time Frame: 16 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: % (value of HbA1c)
Arm/Group | Placebo/KAD-1229 | KAD-1229/KAD-1229
Number analyzed (Participants) | 60 | 118
% (value of HbA1c) | 0.05 (1.04) | -0.61 (0.87)
Statistical Analysis 1: Comparison: Placebo/KAD-1229 vs KAD-1229/KAD-1229; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-0.95 to -0.37]

ADVERSE EVENTS:
Time Frame: Placebo/KAD-1229 and KAD-1229/KAD-1229: 16 weeks, KAD-1229: 52 weeks
Groups:
- Placebo/KAD-1229 (Data Through Week 16): Show the adverse events which occurred with placebo administration during the double-blind period
- KAD-1229/KAD-1229 (Data Through Week 16): Show the adverse events which occurred with KAD-1229 administration during the double-blind period
- KAD-1229 (Data Through Week 52): KDT-1229 administration period in all patients
Arm/Group | Placebo/KAD-1229 (Data Through Week 16) | KAD-1229/KAD-1229 (Data Through Week 16) | KAD-1229 (Data Through Week 52)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/118 | 0/175
Serious Adverse Events (participants affected / at risk) | 2/60 | 4/118 | 18/175
Other Adverse Events (participants affected / at risk) | 19/60 | 28/118 | 98/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/KAD-1229 (Data Through Week 16) (N=60) | KAD-1229/KAD-1229 (Data Through Week 16) (N=118) | KAD-1229 (Data Through Week 52) (N=175)
Pneumonia (Infections and infestations) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 3
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/KAD-1229 (Data Through Week 16) (N=60) | KAD-1229/KAD-1229 (Data Through Week 16) (N=118) | KAD-1229 (Data Through Week 52) (N=175)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 2 | 9 — Corrected as hypoglycaemia
Hunger (General disorders) | 1 | 2 | 9 — Corrected as hypoglycaemia
Asthenia (General disorders) | 2 | 2 | 8 — Corrected as hypoglycaemia
Dizziness (Nervous system disorders) | 1 | 3 | 8 — Corrected as hypoglycaemia
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 6
Palpitations (Cardiac disorders) | 0 | 2 | 6 — Corrected as hypoglycaemia
Nasopharyngitis (Infections and infestations) | 10 | 13 | 49
Bronchitis (Infections and infestations) | 0 | 0 | 6
Headache (Nervous system disorders) | 0 | 2 | 6
Constipation (Gastrointestinal disorders) | 0 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6
Blood triglycerides increased (Investigations) | 1 | 2 | 8
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 6
Tremor (Nervous system disorders) | 1 | 4 | 5 — Corrected as hypoglycaemia
Periodontitis (Infections and infestations) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No